CLINICAL TRIAL: NCT01123824
Title: A Randomized, Double-blind, Double-dummy, Two Period, Two Treatment Cross-over Pharmacodynamic and Pharmacokinetic Study of Clopidogrel Given as 5-day Repeated Oral Doses (300 mg Loading Dose Followed by 75 mg/Day and 600 mg Loading Dose Followed by 150 mg/Day) in 4 Different Groups of CYP2C19 Genotyped Healthy Male and Female Subjects
Brief Title: Pharmacodynamic and Pharmacokinetic Study of 2 Different Dose Regimen of Clopidogrel in CYP2C19 Genotyped Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PKD11147; 2009-010105-37 (EudraCT Number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence clopidogrel 300/75 mg - 600/150 mg (Experimental): Period 1:
  * Day 1: clopidogrel, 300 mg loading dose + placebo
  * Day 2 to Day 5: clopidogrel, 75 mg + placebo, once daily
  Period 2:
  * Day 1: clopidogrel, 600 mg loading dose
  * Day 2 to Day 5: clopidogrel, 150 mg, once daily
  Each intake is at around 8:00 AM fasted for at least 10 hours
  Interventions: Drug: CLOPIDOGREL; Drug: placebo
- Sequence clopidogrel 600/150 mg - 300/75 mg (Experimental): Period 1:
  * Day 1: clopidogrel, 600 mg loading dose
  * Day 2 to Day 5: clopidogrel, 150 mg, once daily
  Period 2:
  * Day 1: clopidogrel, 300 mg loading dose + placebo
  * Day 2 to Day 5: clopidogrel, 75 mg + placebo, once daily
  Each intake is at around 8:00 AM fasted for at least 10 hours
  Interventions: Drug: CLOPIDOGREL; Drug: placebo

INTERVENTIONS:
Drug: CLOPIDOGREL — Pharmaceutical form: tablets
  Route of administration: oral
  Other Names: SR25990
Drug: placebo — Pharmaceutical form: matching tablets
  Route of administration: oral

SUMMARY:
Primary Objective:

* Investigate the possible role of the CYP2C19 genotype in Adenosine diphosphate (ADP)-induced platelet aggregation after administration of a standard dose regimen of clopidogrel (300 mg loading dose followed by 75 mg/day for 4 days) in healthy male and female subjects

Secondary Objectives:

* Assess the pharmacodynamic activity of a higher dose regimen of clopidogrel (600 mg loading dose followed by 150 mg/day for 4 days)
* Compare the pharmacokinetic profiles of clopidogrel active metabolite between the selected groups of genotyped subjects and the 2 dose regimen

DETAILED DESCRIPTION:
The total study duration per subject is 10-12 weeks broken down as follows:

* Screening: 2 to 40 days before the first dosing
* Period 1: 7 days including 5 days treatment
* Washout: At least 14 days after the last dosing
* Period 2: 7 days including 5 days treatment
* End of study: 7 to 10 days after the last dosing

ELIGIBILITY:
Inclusion criteria:

Healthy subject in good health, as determined by a medical history, physical examination including vital signs and clinical laboratory tests:

* with a body weight between 45 kg and 95 kg if male, between 40 kg and 85 kg if female, and with a Body Mass Index (BMI) between 18 and 30 kg/m²
* classified into one of the 4 groups of metabolizers according to his/her CYP2C19 genotype:

  * Ultrarapid Metabolizers (UMs, CYP2C19*1/*17 and CYP2C19*17/*17)
  * homozygous Extensive Metabolizers (homoEMs, CYP2C19*1/*1)
  * heterozygous Extensive Metabolizers (heteroEMs, CYP2C19*1/*2 and CYP2C19*1/*3)
  * Poor Metabolizers (PMs, CYP2C19*2/*2 and CYP2C19*2/*3)

Exclusion criteria:

* Evidence of inherited disorder of coagulation/hemostasis functions
* Subject smoking more than 10 cigarettes or equivalent per day
* Unability to abstain from intake of any drug affecting hemostasis throughout the whole study duration

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maximum platelet aggregation intensity (MAI) induced by Adenosine diphosphate (ADP) 5 µM after 5 days treatment | Day 5 of each period

SECONDARY OUTCOMES:
Maximum platelet aggregation intensity (MAI) induced by ADP 20 µM after 5 days treatment | Day 5 of each period
Platelet reactivity index -Vasodilator-stimulated phosphoprotein test (PRI-VASP) after 5 days treatment | Day 5 of each period
Clopidogrel active metabolite pharmacokinetic parameters (Cmax, tmax, AUC0-24, AUClast) after 5 days treatment | Up to 24 hours postdose on Day 5 for each period

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Study Director, Study Chair — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany

REFERENCES:
- [Result] Simon T, Bhatt DL, Bergougnan L, Farenc C, Pearson K, Perrin L, Vicaut E, Lacreta F, Hurbin F, Dubar M. Genetic polymorphisms and the impact of a higher clopidogrel dose regimen on active metabolite exposure and antiplatelet response in healthy subjects. Clin Pharmacol Ther. 2011 Aug;90(2):287-95. doi: 10.1038/clpt.2011.127. Epub 2011 Jun 29. PMID 21716274